CLINICAL TRIAL: NCT05978700
Title: Effectiveness of Video-game Based Swallowing Function Training in Patients With Dysphagia: a Randomized, Single-blind, Controlled Trial
Brief Title: Effectiveness of Video-game Based Swallowing Function Training in Patients With Dysphagia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ZHANG Bohan (Other)
Responsible Party: Sponsor-Investigator, ZHANG Bohan, Principal Investigator, The Hong Kong Polytechnic University
Organization: The Hong Kong Polytechnic University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HSEARS20230502007
Record Dates: First submitted 2023-07-20; First posted 2023-08-07 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Deglutition Disorders; Rehabilitation; Video Game
MeSH Terms: conditions — Deglutition Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | Unapproved Device: Yes | US Export: No

ARMS (2):
- Video-game group (Experimental): Received the video-game intervention
  Interventions: Device: Video-game
- Conventional therapy group (Active Comparator): Received the conventional therapy intervention
  Interventions: Behavioral: Conventional therapy

INTERVENTIONS:
Device: Video-game — The video-game has three games: (1) Game One - Lip Exercise; (2) Game Two - Tongue Exercises; (3) Game Three - Lower Jaw Exercise. The whole training will take about once a day for 30 min per session, 5 times a week for 4 weeks.
  Arms: Video-game group
Behavioral: Conventional therapy — The control group used the conventional swallowing function training. The lip exercise consisted of the following specific movements: opening mouth, closing mouth, drumming cheeks, left drumming cheeks, and right drumming cheeks; the tongue exercise consisted of the following specific movements: extending the tongue, tongue up, tongue down, tongue left, and tongue right. Each specific movement in the steps lasts 2-3s, repeat 15 times and continue with the next movement. The lower jaw movement contains the following specific movements: keep the head as low as possible, and squeeze the rubber ball placed on the neck for 2-3 seconds, repeat 15 times.
  Arms: Conventional therapy group

SUMMARY:
The goal of this clinical trial is to investigate the effect of video-game on swallowing function in patients with dysphagia through a randomized controlled trial and whether it has additional benefits in improving swallowing function and training compliance compared with conventional training methods. The main questions it aims to answer are:

* How effective is video-game based rehabilitation for dysphagia?
* Whether video-game based has additional benefits in improving swallowing function and training compliance compared with conventional training methods Participants will be divided into two groups, with one group completing video game rehabilitation and one group completing conventional rehabilitation.

ELIGIBILITY:
Inclusion Criteria:

1. first-episode stroke, as confirmed by brain CT or MRI;
2. diagnosis of dysphagia after stroke according to the Toronto Bedside Swallowing Screening Test (TOR-BSST);
3. age between 18 and 80 years;
4. no significant cognitive impairment, able to execute instructions correctly, and with Mini-Mental State Examination (MMSE) score ≥ 24;
5. clear consciousness as assessed by the National Institute of Health stroke scale (NIHSS).

Exclusion Criteria:

1. dysphagia caused by structural lesions (eg, radiotherapy, previous extensive surgery of the head and neck region such as laryngectomy and cordectomy);
2. combined with serious heart, lung, liver, kidney diseases, and hematological disorders;
3. limb deficiency or paralysis, blindness in both eyes, severe visual impairments;
4. motion sickness or vestibular dysfunction;
5. history of epilepsy, malignancy or other neurological diseases;
6. pregnancy or breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2023-10-10 (Actual); Primary Completion 2024-06-01 (Actual); Study Completion 2024-07-31 (Actual)

PRIMARY OUTCOMES:
the Toronto Bedside Swallowing Screening Test (TOR-BSST) | Assessments were conducted at baseline, within 1 week post-training, and week 8.
  The Toronto Bedside Swallowing Screening Test (TOR-BSST) is the best performing water swallow screening tool 8 with a sensitivity of 91.3%, a negative predictive value of 93.3% in the acute phase and 89.5% in the recovery phase. TOR-BSST has shown to be more convenient and cheaper in bedside screening compared to the gold standard method of simultaneous videofluoroscopy (VFSS), which is an invasive assessment. Due to the limitations of the experimental site, the investigators chose TOR-BSST as the assessment tool for dysphagia.
the Functional Oral Intake Scale (FOIS) | Assessments were conducted at baseline, within 1 week post-training, and week 8.
  The Functional Oral Intake Scale consists of a 7-point scale, with level 1 indicating completely impaired oral intake and level 7 indicating complete oral intake regardless of food concentration or type. Scores range from 1 to 7, the higher point means that the participant's oral intake is better.

SECONDARY OUTCOMES:
The swallowing quality of life (SWAL-QOL) questionnaire | Assessments will be conducted at baseline, within 1 week post-training, and week 8.
  The swallowing quality of life (SWAL-QOL) questionnaire consists of 10 subscales and a symptom scale (14 items) to assess the severity of dysphagia symptoms. Scores range from 0 to 100, with lower scores indicating greater impairment of quality of life from dysphagia
The acceptance survey questionnaire | Assessments will be conducted within 1 week post-training.
  The acceptance survey questionnaire was self-designed based on reference to relevant literature, and was repeatedly modified by experts, and consisted of two parts: (1) Basic information: including age, gender, education level, type of work, and disease; (2) Acceptance of video-game based swallowing training: the widely used Technology Acceptance Model (TAM) as a theoretical model , seven dimensions of perceived usefulness, perceived ease of use, perceived ease of learning, perceived applicability, perceived safety, perceived satisfaction, and intension to use, with five questions under each dimension, each scored on a scale of 1 to 5, with 1 being "strongly disagree", 2 being "basically disagree", 3 being "unsure", 4 being "basically agree", and 5 being "strongly agree" , Scores range from 15 to 75, with higher scores indicating that participants are more receptive to video games.
Body mass index (BMI) | Assessments will be conducted at baseline, within 1 week post-training, and week 8.
  Body mass index is one of the most commonly used nutritional assessments among adults.BMI is equal to weight (kg) divided by height (meters squared). Under normal conditions, the BMI is generally between 18 and 24 as normal. When it is lower than 18, it is called underweight; when it is more than 24, it is called overweight; when it is more than 28, it is called obese.
Mini Nutritional Assessment Short Form (MNA-SF) | Assessments will be conducted at baseline, within 1 week post-training, and week 8.
  Mini Nutritional Assessment Short Form (MNA-SF) were used to assess the nutritional status of the dysphagia patients. Scores range from 0 to 14, with >11 identified as malnutrition, ≤11 as normal.
The satisfaction questionnaire | Assessments will be conducted within 1 week post-training.
  The satisfaction questionnaire was designed based on the literatures. There are 15 items, involving 3 dimensions: training mode content setting, training mode format setting, and self-subjective feeling, and scored on a 5-point Likert scale. Scores range from 5 to 15. The higher the score, the more satisfied the patients were with the video-game training.
Adherence | Assessments will be within 1 week post-training.
  Adherence was based on the actual completion of the patient's swallowing function training. The actual completion of the dysphagia training by patients, including the number of training sessions completed and the duration of training, was objectively recorded by the researcher. Adherence was considered good if the patient could complete more than 80% of the training sessions of the corresponding training program; average if the patient could complete 50% to 80% of the training sessions; and poor if the patient could complete less than 50% of the training sessions. Patients are considered to have completed their training when they have completed more than 12 training sessions.
Self-efficacy | Assessments will be conducted at baseline, within 1 week post-training.
  The General Self-Efficacy Scale were used to assess participants' perceptions of learning, with 10 items and scores ranging from 10 to 50, with higher scores indicating higher self-efficacy among participants.
Learned helplessness | Assessments will be conducted at baseline, within 1 week post-training.
  The Learned Helplessness Scale was used to assess participants' feelings of powerlessness over learning, with 18 items and scores ranging from 18 to 90, with higher scores indicating greater powerlessness over learning.

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Xiaotangshan Hospital, Beijing, China, China

IPD SHARING:
Plan to Share IPD: No
Only PI and CI can use IPD.

REFERENCES:
- [Derived] Zhang B, Wong KP, Liu M, Hui V, Guo C, Liu Z, Liu Y, Xiao Q, Qin J. Effect of artificial intelligence-based video-game system on dysphagia in patients with stroke: A randomized controlled trial. Clin Nutr. 2025 Feb;45:81-90. doi: 10.1016/j.clnu.2024.12.022. Epub 2024 Dec 25. PMID 39765160
- [Derived] Zhang B, Wong KP, Liu M, Hui V, Guo C, Liu Y, Liu Z, Liu Y, Xiao Q, Qin J. Face Recognition-Driven Video Game for Dysphagia Rehabilitation in Stroke Patients: A Pilot Randomized Controlled Trial. Arch Phys Med Rehabil. 2025 Mar;106(3):342-350. doi: 10.1016/j.apmr.2024.10.005. Epub 2024 Nov 2. PMID 39491573
- [Derived] Zhang B, Guo C, Hui V, Wong KP, Liu Y, Liu Z, Xu Y, Xiao Q, Chen SC, Qin J. Evaluating the effectiveness of video-game based swallowing function training in patients with dysphagia: study protocol for a randomized controlled trial. Trials. 2023 Nov 16;24(1):735. doi: 10.1186/s13063-023-07738-7. PMID 37974234